CLINICAL TRIAL: NCT02811367
Title: The HPV Self-test as a Test of Cure in the Follow-up of HPV-positive Women in Madagascar
Brief Title: The HPV Self-test as a Test of Cure in Madagascar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Patrick Petignat, Prof., University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-00030
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Human Papilloma Virus Infection; Cervical Intraepithelial Neoplasia Grade 2/3
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus DNA Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV self-test (Experimental): Women will perform the HPV self-test.
  Interventions: Device: HPV test

INTERVENTIONS:
Device: HPV test — Women will perform the HPV self-test and will also undergo a physician-performed HPV test.

SUMMARY:
The purpose of this study is to find out whether Self-HPV may be an accurate method for the follow-up of women with a history of HPV infection.

DETAILED DESCRIPTION:
The efficacy and the availability of cold coagulation render it a valuable technique for the treatment of precancerous lesions in low-resource settings. The Human Papillomavirus (HPV) test performed by women themselves (HPV self-test) could be an efficient method to assess the long-term risk of recurrent/persistent disease in women with a history of HPV infection and cervical intra-epithelial lesions grade 2 or higher (CIN2+).

A total of 443 HPV-positive women, aged 30-65 years, have been selected through a screening campaign conducted in Ambanja, Madagascar, between 2013 and 2015. Of these, 260 have been treated by cold coagulation, conisation or electrocauterization. A follow-up visit at 1-3 years after primary screening will be organized for all HPV-positive women detected at primary screening. Participants will perform an HPV self-test. A sample for cytology and HPV testing will also be collected by the physician. The goal of the study will be the histological search for CIN2+ lesions at one to three years after primary screening.

The investigators expect to see that Self-HPV may be an accurate method for the follow-up of women with a history of HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* women previously positive at HPV testing

Exclusion Criteria:

* pregnancy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cervical intra-epithelial neoplasia grade 2 or worse | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Damien Medical Center, Ambanja, Madagascar, Madagascar

IPD SHARING:
Plan to Share IPD: Undecided